CLINICAL TRIAL: NCT02651376
Title: Safety and Efficacy of Allogenic Adoptive Immune Therapy for Advanced AIDS Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Beijing302H-2
Record Dates: First submitted 2015-09-08; First posted 2016-01-11 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2015-09

CONDITIONS: Human Immunodeficiency Virus; Immunodeficiency
Keywords: Immunodeficiency; Allogenic Mononuclear Cell Transplantation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Immunologic Deficiency Syndromes | interventions — Congresses as Topic; AaIT neurotoxin, Androctonus australis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Conventional plus AAIT (Experimental): Participants received conventional treatment (anti-opportunistic infections and ART) plus a dose (3 times of MNCs) of AAIT.
  Interventions: Combination Product: Conventional plus AAIT

INTERVENTIONS:
Combination Product: Conventional plus AAIT — Participants received conventional (anti-opportunistic infections and ART) treatment and taken i.v., at a roud (3 times) of 2-3*10E8 MNCs/kg body at baseline, week 1 and 2.
  Other Names: Conventional plus allogeneic adoptive immune treatment

SUMMARY:
Combined antiretroviral therapy (cART) efficiently suppress viral replication in majority of AIDS patients. The morbidity and mortality of the disease has dramatically decreased over the past 20 years. However, chronic human immunodeficiency virus-1 (HIV-1) infection lead to profound immune defects in some advanced AIDS patients who often develop with severe opportunistic infections (OIs), severe cachexia and other deadly complications, which accounts for the major death group even under cART. Up-to-date, there are no effective immune interventions to restore host holistic immunity for advanced AIDS patients.

DETAILED DESCRIPTION:
Advanced AIDS patients are usually characterized with CD4 T cells less than 200 cells/uL, including end-stage AIDS patients (CD4 T cells less than 50 cells/uL), and often accompanied with severe opportunistic infections (including tuberculosis, PCP, fungus and so on) and deadly complications.In this regard, advanced AIDS patients present a unique and special profound immune deficiency setting. Therefore, increasing attention and evidence have been paid to development of novel immune therapeutic strategies for those patients.

Immune cell therapy in combination with anti-infection and anti-HIV therapy may open a new direction for advanced AIDS patients, but single cell-based immune therapies do not work well for advanced AIDS patients. Over past 30 years, more than hundreds of AIDS patients with haematological malignancies received autologous or allogeneic hematopoietic stem cell transfusion (HSCT), and their survival rate had been improved to the levels equal to non-HIV patients; however, allogeneic HSCT is only limited to treat AIDS patients with lymphoma or leukemia. The only cured Berlin Patient, who suffered from both acute myeloid leukemia and chronic HIV-1 infection, was transplanted with homozygous CCR5 delta 32 allogeneic HLA-matched stem cells and acquired a long-term remission of both leukemia and AIDS. However, it is very difficult to find the HLA-identical HSCT with CCR5 delta 32 homogenous donors for AIDS patients in clinic. Granulocyte colony-stimulating factor (G-CSF)-mobilized donor peripheral blood mononuclear cells (MNCs) are a heterogeneous population of immune cells that have a potential role in immunomodulation and hemopoiesis. Here, we hypothesized that HLA-mismatched MNCs transfusion can be used to comprehensively restore or boost the host holistic immune system for advanced AIDS patients, to the degree similar as the allogeneic HSCT for leukemia patients.

The purpose of this study is to investigate the safety and initial efficacy of allogeneic adoptive immune therapy (AAIT) for advanced AIDS patients. 20 patients received i.v. transfusion one round (3 times) of 2.0-3.0*10E8 cells/kg of MNSs as the treated group. All of them received the conventional (anti-opportunistic infection and ART) treatment for AIDS. The side effects, symptom improvement, control of opportunistic infections and CD4 T cell numbers will be evaluated during the 48-week follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Severe immunodeficiency patients with chronic HIV-1 infection
2. Advanced patients with CD4 count less than or equal to 200 cells/uL, including end-stage patients with CD4 count less than or equal to 50 cells/uL before entry and at screening
3. With or withour serious complications
4. Ability and willingness to provide informed consent

Exclusion Criteria:

1. Combined with other serious organic diseases, mental illness, including any uncontrolled clinical significance of urinary, respiratory, circulation, nerve, spirit, digestive, endocrine and immune system disease, lymphoma, malignant tumor of blood system etc;
2. Pregnancy, lactation and those who are not pregnant but do not take effective contraceptives measures
3. Allergic to blood products
4. Drug addicts within one year before the test
5. Poor compliance to antiviral therapy; take part in other clinical trials at present, may be contrary to the treatment plan; unable or unwilling to provide informed
6. Other serious conditions that may hamper clinical trials

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Side effects | At Baseline and week 1, 2, 3, 4, 8, 12, 16, 24, 48
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
The changes of clinical symptoms | At Baseline and week 1, 2, 3, 4, 8, 12, 16, 24,48
  Marker for efficacy of treatment
The changes of CD4 T cell counts | At Baseline and week 1, 2, 3, 4, 8, 12, 16, 24, 48
  Marker for host immunity
The plasma RNA copies/mL | At Baseline and at week 4, 12, 24, 48
  Marker for HIV load

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Sheng Wang, Principal Investigator — Beijing 302 Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kuritzkes DR. Hematopoietic stem cell transplantation for HIV cure. J Clin Invest. 2016 Feb;126(2):432-7. doi: 10.1172/JCI80563. Epub 2016 Jan 5. PMID 26731468
- [Background] Hutter G. Stem cell transplantation in strategies for curing HIV/AIDS. AIDS Res Ther. 2016 Sep 13;13(1):31. doi: 10.1186/s12981-016-0114-y. eCollection 2016. PMID 27625700
- [Background] Krishnan A. Stem cell transplantation in HIV-infected patients. Curr Opin HIV AIDS. 2009 Jan;4(1):11-5. doi: 10.1097/COH.0b013e32831a6fc9. PMID 19339935
- [Background] Zhang Z, Fu J, Xu X, Wang S, Xu R, Zhao M, Nie W, Wang X, Zhang J, Li T, Su L, Wang FS. Safety and immunological responses to human mesenchymal stem cell therapy in difficult-to-treat HIV-1-infected patients. AIDS. 2013 May 15;27(8):1283-93. doi: 10.1097/QAD.0b013e32835fab77. PMID 23925377
- [Derived] Yang T, Xie Z, Xu Z, Tu B, Lu H, Huang H, Huang L, Zhang C, Gao L, Jin L, Ma P, Zou J, Liu L, Zhen C, Zhou C, Meng S, Li YY, Song JW, Yang S, Ai HS, Jiao Y, Shi M, Xu R, Wang FS. HLA-mismatched allogeneic adoptive immune therapy in patients with severely immunosuppressed AIDS: a multicenter, open-label, controlled, phase 2a study. Emerg Microbes Infect. 2024 Dec;13(1):2364744. doi: 10.1080/22221751.2024.2364744. Epub 2024 Jun 27. PMID 38935839